CLINICAL TRIAL: NCT02848937
Title: Calcium Mass Balance and Dialytic Efficiency of a New cITRate-containing and Acetate-free Dialysis flUidS: CITRUS Study
Acronym: CITRUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera, Ospedale Civile di Legnano (Other)
Collaborators: AO Garbagnate-Bollate (Unknown)
Responsible Party: Principal Investigator, Carlo Maria Guastoni, DPT Director, Azienda Ospedaliera, Ospedale Civile di Legnano
Other Study IDs: CT-050313
Record Dates: First submitted 2016-07-20; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: ESRD
Keywords: calcium balance; dialysis; concentrate with citrate
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Baths

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bath with citrate: Each patient will participate in two phases of the study. The first phase has the aim to identify the concentration of calcium in the bath with citrate which allows the equivalence of mass balance (Ca_eq) compared to the concentrate with 3 mM acetate and 1.5 mM of calcium (4 weeks). Each week, the concentration of calcium in the bath with citrate is increased from 1.5-, to 1.65, to 1.75 mM.
  •Concentrate SelectBag One (with 3 mM acetic acid) and SelectBag Citrate (with 1 mM of citric acid). The potassium in the bath will be chosen on the basis of the needs of the patient (2 to 3.5 mM) and will be maintained in all concentrates.•All treatment parameters (Qb, time of treatment, weight loss and anticoagulant dose) should be overlapped at all stages of the study
  Interventions: Device: Bath with citrate
- Bath with citrate and Ca_eq: Each patient will participate in two phases of the study. In the second phase will evaluate the effectiveness of the purification concentrate with 1 mM citrate and Ca_eq compared to the concentrate with 3 mM acetate and 1.5 mM calcium. For each of the sessions will be used the following materials:
  * Filter high permeability (Kuf> 20ml/mmHg);
  * Concentrate SelectBag One (with 3 mM acetic acid) and SelectBag Citrate (with 1 mM of citric acid). The potassium in the bath will be chosen on the basis of the needs of the patient (2 to 3.5 mM) and will be maintained in all concentrates.
  * All treatment parameters (Qb, time of treatment, weight loss and anticoagulant dose) should be overlapped at all stages of the study.
  Interventions: Device: Bath with citrate and Ca_eq

INTERVENTIONS:
Device: Bath with citrate — bath with citrate which allows the equivalence of mass balance (Ca_eq) compared to the concentrate with 3 mM acetate and 1.5 mM of calcium
  Other Names: Select Bag Citrate
  Groups: Bath with citrate
Device: Bath with citrate and Ca_eq — bath with citrate and Ca_eq of concentrate with 3 mM acetate and 1.5 mM of calcium
  Other Names: Select Bag Citrate
  Groups: Bath with citrate and Ca_eq

SUMMARY:
This study aimed to evaluate the effect on the calcium balance of a concentrate with 1 mM citrate and locate the equivalent concentration of calcium (Ca_eq) at a concentration of 3 mM acetate and traditional with 1.5 mM calcium in HD. The secondary objective is to evaluate the performance in the medium term of purifying the concentrate with 1 mM citrate and Ca_eq, compared to traditional concentrated with 3 mM acetate and 1.5 mM calcium in HD.

DETAILED DESCRIPTION:
Primary Objective The primary objective of this study is to find the formulation of calcium (1.50, 1.65 and 1.75 mM) in the bath with 1 mM citrate which allows the equivalence of calcium balance (Ca_eq) in a sitting HD compared to traditional concentrated with 3 mM of calcium acetate and 1.5.

Secondary objectives

* Evaluate the purifying performance of small and medium-sized molecules in HD with concentrated with 1 mM citrate and Ca_eq compared to traditional concentrated with 3 mM calcium acetate and 1.5.
* Observe the effects on hemodynamic of the concentrate through the variation of the pre and post-dialysis blood pressure and intradialytic symptoms (cramps, hypotension, headache).
* Evaluate the variations of the parameters of mineral metabolism: Predialytic values of PTH, alkaline phosphatase treatments with concentrated Cit (1 mM citrate and Ca_eq) and concentrated with traditional Ac (3 mM calcium acetate and 1.5).

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically stable.

  * age> 18 years.
  * HD therapy for more than 3 months.
  * good vascular access native functionality that enables real blood flow of at least 250 ml / min.

Exclusion Criteria:

* Patients with the features listed below may not be enrolled in this survey:

  * Life expectancy <6 months.
  * residual diuresis> 500 ml / day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients clinically stable.
  * age> 18 years.
  * HD therapy for more than 3 months.
  * good vascular access native functionality that enables real blood flow of at least 250 ml / min.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Plasma calcium level evaluation (mEq/l) | 6 months
  Calcium balance from data of the calcium ion and total dialysate compartment. Complete blood count pre-and post-dialysis, total Proteins pre-and post-dialysis, will be collected from the patient's blood sitting in the middle of the week. Biochemical data from the dialysis fluid and spent dialysate sitting in the middle of the week:Calcium ion (EGA) and total in the dialysis fluid in the following times: 5, 120, end of dialysis; Calcium ion (EGA) and total effluent in the following times: 5, 120, end of dialysis

SECONDARY OUTCOMES:
Evaluate purifying performance of small and medium-sized molecules in HD (Kt/V) | 6 months
  Evaluate the purifying performance of small and medium-sized molecules in HD (EKt/V) with concentrated with 1 mM citrate and Ca_eq compared to traditional concentrated with 3 mM calcium acetate and 1.5
Evaluation of variations of the parameters of mineral metabolism | 6 months
  Evaluate the variations of the parameters of mineral metabolism: Predialytic values of PTH (mEq/l), alkaline phosphatase treatments (U/I) with concentrated Cit (1 mM citrate and Ca_eq) and concentrated with traditional Ac (3 mM calcium acetate and 1.5

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Maria Guastoni, DR, Principal Investigator — Asst Ovest Mi
Locations (1):
- Carlo Maria Guastoni, Legnano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahmad S, Callan R, Cole JJ, Blagg CR. Dialysate made from dry chemicals using citric acid increases dialysis dose. Am J Kidney Dis. 2000 Mar;35(3):493-9. doi: 10.1016/s0272-6386(00)70203-4. PMID 10692276
- [Background] Bauer E, Derfler K, Joukhadar C, Druml W. Citrate kinetics in patients receiving long-term hemodialysis therapy. Am J Kidney Dis. 2005 Nov;46(5):903-7. doi: 10.1053/j.ajkd.2005.07.041. PMID 16253731
- [Background] Kossmann RJ, Gonzales A, Callan R, Ahmad S. Increased efficiency of hemodialysis with citrate dialysate: a prospective controlled study. Clin J Am Soc Nephrol. 2009 Sep;4(9):1459-64. doi: 10.2215/CJN.02590409. Epub 2009 Aug 6. PMID 19661218
- [Background] Bosticardo G, Malberti F, Basile C, Leardini L, Libutti P, Filiberti O, Schillaci E, Ravani P. Optimizing the dialysate calcium concentration in bicarbonate haemodialysis. Nephrol Dial Transplant. 2012 Jun;27(6):2489-96. doi: 10.1093/ndt/gfr733. Epub 2012 Feb 21. PMID 22357700